CLINICAL TRIAL: NCT01618708
Title: A Pivotal, Multicenter, Double Blind Study of the Safety and Effectiveness of Synvisc-One® (Hylan G-F 20) in Patients With Mild to Moderate Primary Osteoarthritis of the Hip
Brief Title: A Study of the Safety and Effectiveness of Synvisc-One® (Hylan G-F 20) in Patients With Primary Osteoarthritis of the Hip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SYNV04910; EFC12791 (Other: Sanofi)
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-05

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Synvisc-One (Experimental): Single intraarticular (IA) injection of Synvisc-One (48 mg of Hylan G-F 20 polymer) at Day 1. Participants were observed for 26 weeks in follow up period.
  Interventions: Device: Synvisc-One (hylan G-F 20)
- Placebo (Placebo Comparator): Single IA injection of placebo matched to Synvisc-One at Day 1. Participants were observed for 26 weeks in follow up period.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Synvisc-One (hylan G-F 20) — 6-mL IA injection
  Arms: Synvisc-One
Device: Placebo — 6 mL injection of phosphate buffered saline
  Arms: Placebo

SUMMARY:
The primary objective of this study was to demonstrate any changes in assessments of pain for participants receiving Synvisc-One compared to control.

ELIGIBILITY:
Inclusion Criteria:

* The participant had symptomatic osteoarthritis (OA) in the target joint
* The participant had a diagnosis of primary OA of the hip at Screening according to the American College of Rheumatology (ACR) Criteria
* The participant, if female and of childbearing potential, must had a negative pregnancy test and had taken oral contraceptives for at least 1 month prior to treatment and continued for the duration of the study (up to and including the final study visit), or agreed to use 2 forms of contraception (e.g., condoms plus spermatocide), otherwise females must be surgically sterile, or postmenopausal for at least 1 year

Exclusion Criteria:

* The participant had symptomatic OA in the contralateral hip with a Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) A1 numerical rating scale (NRS) score of ≥ 4 at Screening (symptomatic OA with a WOMAC A1 NRS score of 0-3 in the contralateral hip was allowed)
* The participant if a woman was pregnant, lactating, or unwilling to use adequate contraception
* The participant had prior viscosupplementation therapy in the target hip joint within 26 weeks of Screening
* The participant had a known history of hypersensitivity to avian protein or any components of hyaluronan-based injection devices
* The participant had a known history of hypersensitivity to steroids, lidocaine, and/or acetaminophen
* The participant had a known history of hypersensitivity to injected contrast agent at a previous radiological examination (e.g., computed tomography [CT] scan, angiogram, etc.), or known history of hypersensitivity to shellfish or iodine, or any other impediment to the hip injection procedure
* The participant had active infection in the area of the injection site
* The participant had any major surgery, arthroplasty or arthroscopy in the target hip or lower extremities within 26 weeks of Screening, or planned surgery in the lower extremities throughout the duration of the study infectious complications
* The participant used an investigational drug, device or biologic within 12 weeks of Screening
* The participant had any significant medical condition that the Investigator feels would interfere with study evaluations and study participation

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2012-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (48):
- United States (45):
  - Investigational Site Number 840025, Burmingham, Alabama
  - Investigational Site Number 840042, Phoenix, Arizona
  - Investigational Site Number 840056, Phoenix, Arizona
  - Investigational Site Number 840004, Tucson, Arizona
  - Investigational Site Number 840023, Covina, California
  - Investigational Site Number 840058, La Mesa, California
  - Investigational Site Number 840022, Santa Monica, California
  - Investigational Site Number 840050, Farmington, Connecticut
  - Investigational Site Number 840027, Stamford, Connecticut
  - Investigational Site Number 840051, Waterbury, Connecticut
  - Investigational Site Number 840011, Bradenton, Florida
  - Investigational Site Number 840036, Fort Lauderdale, Florida
  - Investigational Site Number 840017, Jupiter, Florida
  - Investigational Site Number 840038, New Port Richey, Florida
  - Investigational Site Number 840041, Pensacola, Florida
  - Investigational Site Number 840047, Sarasota, Florida
  - Investigational Site Number 840049, South Miami, Florida
  - Investigational Site Number 840039, Marietta, Georgia
  - Investigational Site Number 840005, Meridian, Idaho
  - Investigational Site Number 840002, Chicago, Illinois
  - Investigational Site Number 840043, Wichita, Kansas
  - Investigational Site Number 840012, Lexington, Kentucky
  - Investigational Site Number 840033, Traverse City, Michigan
  - Investigational Site Number 840037, St Louis, Missouri
  - Investigational Site Number 840007, Reno, Nevada
  - Investigational Site Number 840048, Egg Harbor, New Jersey
  - Investigational Site Number 840024, Amherst, New York
  - Investigational Site Number 840029, Hartsdale, New York
  - Investigational Site Number 840014, Rochester, New York
  - Investigational Site Number 840044, Asheville, North Carolina
  - Investigational Site Number 840028, Raleigh, North Carolina
  - Investigational Site Number 840045, Wilmington, North Carolina
  - Investigational Site Number 840046, Columbus, Ohio
  - Investigational Site Number 840013, Altoona, Pennsylvania
  - Investigational Site Number 840055, Philadelphia, Pennsylvania
  - Investigational Site Number 840018, Reading, Pennsylvania
  - Investigational Site Number 840026, Mt. Pleasant, South Carolina
  - Investigational Site Number 840052, Memphis, Tennessee
  - Investigational Site Number 840054, Austin, Texas
  - Investigational Site Number 840040, Bedford, Texas
  - Investigational Site Number 840010, Dallas, Texas
  - Investigational Site Number 840009, Draper, Utah
  - Investigational Site Number 840032, Salt Lake City, Utah
  - Investigational Site Number 840016, Charlottesville, Virginia
  - Investigational Site Number 840003, Seattle, Washington
- Canada (3):
  - Investigational Site Number 124091, London
  - Investigational Site Number 124093, Montreal
  - Investigational Site Number 124092, Sherbrooke

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 42 centers in the US and Canada. A total of 1113 participants were screened between 05 September 2012 and 21 November 2014.
Pre-assignment Details: Of 1113 screened participants, 33 were re-screened, 357 were randomized and 741 were screen failures. Screen failures were mainly due to inclusion criteria not met and exclusion criteria met.
Groups:
- Placebo: Single 6 mL intraarticular (IA) injection of placebo matched to Synvisc-One (phosphate buffered saline) at Day 1. Participants were observed for 26 weeks in follow up period.
- Synvisc-One: Single 6 mL IA injection of Synvisc-One (48 mg of Hylan G-F 20 polymer) at Day 1. Participants were observed for 26 weeks in follow up period.
Period: Overall Study
Arm/Group | Placebo | Synvisc-One
Started | 175 | 182
Treated | 172 | 180
Completed | 131 | 136
Not Completed | 44 | 46
Not completed — Adverse Event | 10 | 10
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 17 | 22
Not completed — Lack of Efficacy | 8 | 8
Not completed — Technical problems | 2 | 0
Not completed — Other than specified above | 1 | 1
Not completed — Randomized but not treated | 3 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants who received study medication or part of the treatment administration.
Groups:
- Placebo: Single 6 mL IA injection of placebo matched to Synvisc-One (phosphate buffered saline) at Day 1. Participants were observed for 26 weeks in follow up period.
- Total: Total of all reporting groups
Arm/Group | Placebo | Synvisc-One | Total
Number analyzed (Participants) | 175 | 182 | 357
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (8.8) | 60.8 (10.0) | 60.3 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 106 | 211
  Male | 70 | 76 | 146

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) A1 Subscore (Walking Pain) Over 26 Weeks
Description: WOMAC Numerical Rating Scale (NRS) 3.1 questionnaire is a health status measure questionnaire of 24 questions comprising 3 subscales (pain, stiffness and physical function). WOMAC A1 (measure of pain during walking on a flat surface) was measured on 11-point (NRS) ranging from 0 (none) to 10 (extreme), where lower score represents lower pain and higher score represents higher pain.
Time Frame: From baseline to Week 26
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Synvisc-One
Number analyzed (Participants) | 175 | 182
units on a scale | -2.26 (0.17) | -2.19 (0.16)
Statistical Analysis 1: Comparison: Placebo vs Synvisc-One; Synvisc-One group was compared to placebo group using mixed model for repeated measures (MMRM) approach assuming missing data at random (MAR); Test type: Superiority or Other; p = 0.7462, Mixed Models Analysis — Threshold for significance at 0.05 level; Least Squares (LS) Mean difference = 0.07, 95% CI 2-sided [-0.38 to 0.52] — Placebo vs Synvisc-One

2. Secondary Outcome: Change From Baseline in WOMAC A Score Over 26 Weeks
Description: WOMAC NRS 3.1 questionnaire is a health status measure questionnaire of 24 questions comprising 3 subscales (pain, stiffness and physical function). WOMAC A (measure of pain) was measured on 11-point NRS ranging from 0 (none) to 10 (extreme), where lower score represents lower pain and higher score represents higher pain.
Time Frame: From Baseline to Week 26
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Single 6 mL IA injection of placebo matched to Synvisc-One at Day 1. Participants were observed for 26 weeks in follow up period.
Arm/Group | Placebo | Synvisc-One
Number analyzed (Participants) | 175 | 182
units on a scale | -2.26 (0.16) | -2.19 (0.16)

3. Secondary Outcome: Change From Baseline in Patient Global Self-Assessment (PTGA) Score Over 26 Weeks
Description: PTGA (self-assessment of target hip osteoarthritis condition) was measured using the 11-point NRS ranging from 0 (none) to 10 (extreme), where lower score represents very well condition and higher score represents very poor condition.
Time Frame: From baseline to Week 26
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Synvisc-One
Number analyzed (Participants) | 175 | 182
units on a scale | -2.06 (0.17) | -2.00 (0.16)

4. Secondary Outcome: Percentage of WOMAC A1 Responder Over 26 Weeks
Description: WOMAC A1 responder rate defined as ≥2 point improvement on 11-point NRS Scale, generalized estimating equations modeling was used for the analysis of WOMAC A1 responders.
Time Frame: From Baseline to Week 26
Population: ITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Synvisc-One
Number analyzed (Participants) | 175 | 182
Percentage of participants | 45.71 | 45.05

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 26) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is any AE that started during or after the first dose of study drug. Safety population defined as all randomized participants who received any study drug or part of treatment administration.
Arm/Group | Placebo | Synvisc-One
Serious Adverse Events (participants affected / at risk) | 15/172 | 10/180
Other Adverse Events (participants affected / at risk) | 33/172 | 43/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=172) | Synvisc-One (N=180)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Intracranial lipoma (Congenital, familial and genetic disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obesity surgery (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=172) | Synvisc-One (N=180)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 32
Headache (Nervous system disorders) | 14 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.